CLINICAL TRIAL: NCT01570374
Title: Internet-based Treatment of Generalized Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Per Carlbring, PhD, Professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Oroshjalpen
Record Dates: First submitted 2012-03-31; First posted 2012-04-04 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Generalized Anxiety Disorder
Keywords: Cognitive behavioral therapy; Internet; Anxiety; Generalized anxiety disorder
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- iCBT (Experimental): Receives treatment.
  Interventions: Behavioral: Internet-based cognitive behavioral therapy (iCBT)
- Waiting list control group (No Intervention): The waiting list control group initially receives no treatment, but do weekly screenings. After 9 weeks, the control group receives the same treatment as the other study arm.

INTERVENTIONS:
Behavioral: Internet-based cognitive behavioral therapy (iCBT) — 9 week internet-administered, therapist-assisted, controlled-progression cognitive behavioral therapy (iCBT). Individualized and disorder-specific.
  Arms: iCBT

SUMMARY:
The purpose of this study is to determine whether internet-administered cognitive behavior therapy is a feasible treatment for generalized anxiety disorder.

ELIGIBILITY:
Inclusion Criteria:

* Satisfy DSM-IV criteria for generalized anxiety disorder
* Living in Sweden and being able to read Swedish
* Access to computer with internet connection

Exclusion Criteria:

* Currently receiving other psychological treatment
* Non-stable use of psychoactive medication
* Deemed suicidal
* Deemed to suffer from other psychological disorder, e.g. psychosis, bipolarity etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2012-01; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Penn State Worry Questionnaire (PSWQ) | 24 hours
  Measures anxiety symptoms related to Generalized Anxiety Disorder. 16 items.
Change from baseline in Penn State Worry Questionnaire (PSWQ) | 6 months
  Measures anxiety symptoms related to Generalized Anxiety Disorder. 16 items.
Change from baseline in Penn State Worry Questionnaire (PSWQ) | 12 months
  Measures anxiety symptoms related to Generalized Anxiety Disorder. 16 items.
Change from baseline in Penn State Worry Questionnaire (PSWQ) | 24 months
  Measures anxiety symptoms related to Generalized Anxiety Disorder. 16 items.

SECONDARY OUTCOMES:
Change from baseline in Beck Anxiety Inventory (BAI) | 24 hours
  21 item rating scale for anxiety symptoms.
Change from baseline in Beck Anxiety Inventory (BAI) | 6 months
  21 item rating scale for anxiety symptoms.
Change from baseline in Beck Anxiety Inventory (BAI) | 12 months
  21 item rating scale for anxiety symptoms.
Change from baseline in Beck Anxiety Inventory (BAI) | 24 months
  21 item rating scale for anxiety symptoms.
Change from baseline in Quality Of Life Inventory (QOLI) | 24 hours
  The QOLI assessment yields an overall score and a profile of problems and strengths in 16 areas of life such as love, work and play. The QOLI test is a measure of positive psychology and positive mental health.
Change from baseline in Quality Of Life Inventory (QOLI) | 6 months
  The QOLI assessment yields an overall score and a profile of problems and strengths in 16 areas of life such as love, work and play. The QOLI test is a measure of positive psychology and positive mental health.
Change from baseline in Quality Of Life Inventory (QOLI) | 12 months
  The QOLI assessment yields an overall score and a profile of problems and strengths in 16 areas of life such as love, work and play. The QOLI test is a measure of positive psychology and positive mental health.
Change from baseline in Quality Of Life Inventory (QOLI) | 24 months
  The QOLI assessment yields an overall score and a profile of problems and strengths in 16 areas of life such as love, work and play. The QOLI test is a measure of positive psychology and positive mental health.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | 24 hours
  9-item depression rating scale.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | 6 months
  9-item depression rating scale.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | 12 months
  9-item depression rating scale.
Change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) | 24 months
  9-item depression rating scale.
Change from baseline in Patient Health Questionnaire (PHQ-9) | Weekly during treatment period
  The PHQ-9 is the nine item depression scale of the Patient Health Questionnaire. The PHQ-9 is a powerful tool for assisting primary care clinicians in diagnosing depression as well as selecting and monitoring treatment. The PHQ-9 is based directly on the diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual Fourth Edition (DSM-IV).
Change from baseline in Patient Health Questionnaire (PHQ-9) | 24 hours
  The PHQ-9 is the nine item depression scale of the Patient Health Questionnaire. The PHQ-9 is a powerful tool for assisting primary care clinicians in diagnosing depression as well as selecting and monitoring treatment. The PHQ-9 is based directly on the diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual Fourth Edition (DSM-IV).
Change from baseline in Patient Health Questionnaire (PHQ-9) | 6 months
  The PHQ-9 is the nine item depression scale of the Patient Health Questionnaire. The PHQ-9 is a powerful tool for assisting primary care clinicians in diagnosing depression as well as selecting and monitoring treatment. The PHQ-9 is based directly on the diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual Fourth Edition (DSM-IV).
Change from baseline in Patient Health Questionnaire (PHQ-9) | 12 months
  The PHQ-9 is the nine item depression scale of the Patient Health Questionnaire. The PHQ-9 is a powerful tool for assisting primary care clinicians in diagnosing depression as well as selecting and monitoring treatment. The PHQ-9 is based directly on the diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual Fourth Edition (DSM-IV).
Change from baseline in Patient Health Questionnaire (PHQ-9) | 24 months
  The PHQ-9 is the nine item depression scale of the Patient Health Questionnaire. The PHQ-9 is a powerful tool for assisting primary care clinicians in diagnosing depression as well as selecting and monitoring treatment. The PHQ-9 is based directly on the diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual Fourth Edition (DSM-IV).
Change from baseline in Generalized Anxiety Disorder-7 (GAD-7) | Weekly during treatment period
  7-item screening form for Generalized Anxiety Disorder.
Change from baseline in Generalized Anxiety Disorder-7 (GAD-7) | 24 hours
  7-item screening form for Generalized Anxiety Disorder.
Change from baseline in Generalized Anxiety Disorder-7 (GAD-7) | 6 months
  7-item screening form for Generalized Anxiety Disorder.
Change from baseline in Generalized Anxiety Disorder-7 (GAD-7) | 12 months
  7-item screening form for Generalized Anxiety Disorder.
Change from baseline in Generalized Anxiety Disorder-7 (GAD-7) | 24 months
  7-item screening form for Generalized Anxiety Disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Per Carlbring, Professor, Principal Investigator — Department of Psychology, Umeå University
Locations (1):
- Department of Psychology, Umeå University, Umeå, Västerbotten County, Sweden

REFERENCES:
- [Result] Dahlin M, Andersson G, Magnusson K, Johansson T, Sjogren J, Hakansson A, Pettersson M, Kadowaki A, Cuijpers P, Carlbring P. Internet-delivered acceptance-based behaviour therapy for generalized anxiety disorder: A randomized controlled trial. Behav Res Ther. 2016 Feb;77:86-95. doi: 10.1016/j.brat.2015.12.007. Epub 2015 Dec 21. PMID 26731173